CLINICAL TRIAL: NCT00185666
Title: Cyberknife Precision Radiation Delivery System for Tumors of the Spine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Iris Catrice Gibbs, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPN0001; NCT00185666; SPN0001
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Spinal Cord Cancer; Brain (Nervous System) Cancers
MeSH Terms: conditions — Neurologic Manifestations; Neoplasms | interventions — Radiosurgery

INTERVENTIONS:
Procedure: Stereotactic radiosurgery

SUMMARY:
The purpose of this study is to determine the usefulness of Cyberknife precision radiation in eliminating or preventing the further growth of spinal tumors and lesions.

ELIGIBILITY:
Inclusion Criteria:- Intra-axial, extra-axial, or vertebral spinal lesion

* Age > 5
* Histologic confirmation of malignant primary lesion or radiographic diagnosis of benign or vascular spinal lesion
* No rapidly deteriorating symptoms of spinal cord compression
* No instability of the spine
* Life expectancy > 6 months Exclusion Criteria:- Patients without tumors of the spine
* Patients younger than 5 years old

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Usefulness of Cyberknife precision radiation in eliminating or preventing the further growth of spinal tumors and lesions | completed

CONTACTS AND LOCATIONS:
Overall Officials: Iris Catrice Gibbs, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Gibbs IC, Chang SD. Radiosurgery and radiotherapy for sacral tumors. Neurosurg Focus. 2003 Aug 15;15(2):E8. doi: 10.3171/foc.2003.15.2.8. PMID 15350039
- [Result] Gibbs IC, Kamnerdsupaphon P, Ryu MR, Dodd R, Kiernan M, Chang SD, Adler JR Jr. Image-guided robotic radiosurgery for spinal metastases. Radiother Oncol. 2007 Feb;82(2):185-90. doi: 10.1016/j.radonc.2006.11.023. Epub 2007 Jan 24. PMID 17257702
- [Result] Dodd RL, Ryu MR, Kamnerdsupaphon P, Gibbs IC, Chang SD Jr, Adler JR Jr. CyberKnife radiosurgery for benign intradural extramedullary spinal tumors. Neurosurgery. 2006 Apr;58(4):674-85; discussion 674-85. doi: 10.1227/01.NEU.0000204128.84742.8F. PMID 16575331
- [Result] Sinclair J, Chang SD, Gibbs IC, Adler JR Jr. Multisession CyberKnife radiosurgery for intramedullary spinal cord arteriovenous malformations. Neurosurgery. 2006 Jun;58(6):1081-9; discussion 1081-9. doi: 10.1227/01.NEU.0000215891.25153.BA. PMID 16723887